CLINICAL TRIAL: NCT04015700
Title: A Pilot Study to Assess the Safety, Feasibility, and Immunogenicity of a Neoantigen-based Personalized in Patients With Newly Diagnosed, Unmethylated Glioblastoma
Brief Title: Neoantigen-based Personalized DNA Vaccine in Patients With Newly Diagnosed, Unmethylated Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Geneos Therapeutics (Industry); The Foundation for Barnes-Jewish Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202003072; R01NS112712 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Vaccines; rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vaccine (GNOS-PV01 + INO-9012) (Experimental): * Standard radiation therapy will be administered per standard of care and is outside the scope of this study.
  * GNOS-PV01 + INO-9012 will be given on Days 1, 22, and 43 of Cycle 1 and then on Day 1 of each subsequent cycle beginning with Cycle 2.
  Interventions: Biological: Personalized neoantigen DNA vaccine supplied by Geneos Therapeutics; Device: CELLECTRA®2000 EP Device supplied by Geneos Therapeutics; Drug: Plasmid encoded IL-12

INTERVENTIONS:
Biological: Personalized neoantigen DNA vaccine supplied by Geneos Therapeutics — -The neoantigen DNA vaccines are also known as DNA plasmid vector expressing tumor-specific antigens.
  Other Names: GNOS-PV01; Vaccine
Device: CELLECTRA®2000 EP Device supplied by Geneos Therapeutics — CELLECTRA® 2000 Device is a system indicated for use to enhance the uptake and expression of plasmid-based biologics in order to enhance vaccine efficacy.
Drug: Plasmid encoded IL-12 — The INO-9012 vials will be supplied by Geneos Therapeutics
  Other Names: INO-9012

SUMMARY:
This is a single institution, open-label, single arm, study assessing the safety, feasibility, and immunogenicity of a personalized neoantigen-based vaccine in subjects with newly diagnosed, unmethylated glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically confirmed MGMT unmethylated glioblastoma multiforme (WHO grade IV). Patients with secondary glioblastoma, in particular those who are IDH1 or IDH2 mutant, will not be excluded. High grade gliomas with molecular features of glioblastoma will be included. MGMT methylation status must be confirmed by standard a PCR-based assay.
* Patients who had prior craniotomy with biopsy, subtotal resection, total gross resection, or re-resection will be permitted.
* Consent to genome sequencing and dbGaP-based data sharing and has provided or will provide germline (PBMC) and tumor DNA/RNA samples of adequate quality for sequencing. (Acquisition of specimens for sequencing and the sequencing itself may be done as part of routine care or another research project.)
* At least 18 years of age.
* Karnofsky performance status ≥ 60%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Systemic corticosteroid therapy is permitted provided dosing is no greater than 4 mg per day (dexamethasone or equivalent) on the day of vaccine administration.
* Bevacizumab will be allowed if given for symptomatic control of vasogenic edema and to avoid high dose of corticosteroids.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation, including at least 5 months (for women of childbearing potential) and at least 7 months (for men) after last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* As this study aims to assess the immunogenicity of personalized neoantigen DNA vaccine plus plasmid encoded IL-12 as an adjuvant, no prior immunotherapy will be permitted.
* Inadequate tissue acquisition to allow for neoantigen screening.
* No candidate neoantigen identified during screening.
* A history of other malignancy ≤ 3 years previous with the exception of non-melanoma skin cancer, any in situ cancer that has been successfully resected and cured, treated superficial bladder cancer, or any early-stage solid tumor that was successfully resected without need for adjuvant radiation or chemotherapy.
* Receiving any other investigational agents within 4 weeks of beginning study treatment.
* Known allergy, or history of serious adverse reaction to, vaccines such as anaphylaxis, hives, or respiratory difficulty.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to any agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of immunodeficiency disorder or autoimmune condition requiring active immunosuppressive therapy. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines.
* Presence of clinically significant increased intracranial pressure (e.g. impending herniation) or hemorrhage, uncontrolled seizures, or requirement for immediate palliative treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of first dose of vaccine.
* Presence of acute or chronic bleeding or clotting disorder that would contraindicate IM injections
* Fewer than 2 acceptable sites available for IM injection and CELLECTRA® 2000 EP considering the deltoid and anterolateral quadriceps muscles:

  * Tattoos, keloids, or hypertrophic scars located within 2 cm of intended administration site
  * Implantable-cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the deltoid injection site (unless deemed acceptable by a cardiologist)
  * Any metal implants or implantable medical device within the intended treatment site (i.e. electroporation area).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2027-09-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a personalized neoantigen DNA vaccine as measured by dose-limiting toxicities (DLTs) | Up to 30 days
  A DLT will be defined as any grade 3 toxicity or greater according to CTCAE v5 considered at least possibly related to study treatment. The DLT observation period begins with Cycle 1 Day 1 (date of first vaccine administration) and continues for 30 days
Feasibility of generating a personalized neoantigen DNA vaccine for patients with newly diagnosed, unmethylated GBM as measured by the ability to identify candidate tumor-specific neoantigens | 4 weeks post-completion of radiotherapy (day 1 of treatment regimen)
Feasibility of generating a personalized neoantigen DNA vaccine for patients with newly diagnosed, unmethylated GBM as measured by the ability to manufacture a neoantigen-based DNA vaccine | 4 weeks post-completion of radiotherapy (day 1 of treatment regimen)
Feasibility of generating a personalized neoantigen DNA vaccine for patients with newly diagnosed, unmethylated GBM as measured by the ability to administer the vaccine to a patient | 4 weeks post-completion of radiotherapy (day 1 of treatment regimen)

SECONDARY OUTCOMES:
Immunogenicity of a personalized neoantigen DNA vaccine as measured by the ability to generate a measurable neoantigen-specific CD8 T cell response in vaccinated patients | Week 10 post-vaccination
Immunogenicity of a personalized neoantigen DNA vaccine as measured by the number of individual neoantigens per number of neoantigens vaccinated against, with which a measurable CD8 T cell-specific response is identified | Week 10 post-vaccination
Number of high quality candidates neoantigens present in patients with newly diagnosed GBM | Week 24 post-vaccination
  -High quality neoantigens will be defined as those that meet criteria for inclusion in a vaccine
Progression-free survival (PFS) rate | 6 months
  * PFS=duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progression: any of the following
    * ≥ 25% increase in sum products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline or best response, on stable or increasing doses of corticosteroids*. The absolute increase in any dimension must be at least 5mm when calculating the products.
    * Significant increase in T2/FLAIR nonenhancing lesion on stable/increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy* not caused by comorbid events
    * New measureable lesion.
    * Clear clinical deterioration not attributable to other causes apart from the tumor (e.g. seizures, medication adverse effects, complications of therapy, cerebrovascular events, infection, and so on) or changes in corticosteroid dose.
Overall survival rate | 12 months
Immunogenicity of a personalized neoantigen DNA vaccine as measured by T-cell phenotype, myeloid derived suppressor cell frequency by flow cytometry | Week 24 post-vaccination
Immunogenicity of a personalized neoantigen DNA vaccine as measured by diversity of clonality from T cell receptor sequencing | Week 24 post-vaccination
Immunogenicity of a personalized neoantigen DNA vaccine as measured by putative antigen specificity from T cell receptor sequencing | Week 24 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tanner M Johanns, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu